CLINICAL TRIAL: NCT00271687
Title: A Pilot Study of Exercise in Patients With Docetaxel-Based Chemotherapy for Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-14-0049 / 22262
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Prostatic Neoplasms; Neoplasm Metastasis; Palliative Care
Keywords: exercise; exercise therapy; activities of daily living; quality of life
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Exercise training

SUMMARY:
This study aims to provide preliminary data on the feasibility and outcomes of a 12 week exercise program on the quality of life of men with hormone refractory prostate cancer receiving docetaxel-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of prostate cancer
* receiving docetaxel-based chemotherapy at the CCI
* age 18 years or over
* approval of oncologist
* informed written consent

Exclusion Criteria:

* life expectancy less than 6 months
* Karnofsky performance score less than 70
* contraindications for exercise (e.g. uncontrolled cardiac, respiratory, hypertensive or psychiatric disorder)
* unable to understand, read, write and speak English
* unable or unwilling to attend supervised exercise sessions 3 times weekly
* unable or unwilling to complete outcome assessments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
feasibility (recruitment, adherence, safety)

SECONDARY OUTCOMES:
quality of life
functional abilities

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Courneya, M.D., Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada